CLINICAL TRIAL: NCT06775028
Title: AFFIRMO - Atrial Fibrillation Integrated Approach in Frail, Multimorbid and Polymedicated Older People
Brief Title: Integrated Approach in Frail Older People with Atrial Fibrillation
Acronym: AFFIRMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Care Foundation (Other)
Collaborators: Aalborg University (Other); University of Belgrade (Other); Universidad de Murcia (Other); Carol Davila University of Medicine and Pharmacy (Other); Plovdiv Medical University (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23
Record Dates: First submitted 2024-12-31; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF); Hypertension; Coronary Arterial Disease (CAD); Heart Failure; COPD; Peripheral Arterial Disease; CKD; Diabetes Mellitus; Stroke; TIA (Transient Ischemic Attack)
Keywords: iABC; Atrial Fibrillation; Cluster Trial
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Heart Failure; Pulmonary Disease, Chronic Obstructive; Peripheral Arterial Disease; Diabetes Mellitus; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quality-improvement intervention (iABC) (Experimental): The novel platform (iABC) that will be used in AFFIRMO will consist of an educational program, a healthy or functional diet/physical activity, guideline-adherent drug treatments, periodic (re)assessment.
  iABC will provide guidance to obtain a more personalized care to AF patients in the experimental cluster implementing specific strategies to obtain clinical control for all the three pillars of the ABC pathway. During the entire follow-up the physician will be able to check the data imputed by the patients and, eventually, contact the patient to provide recommendations and to discuss changes to the treatments and lifestyle habits.
  Interventions: Other: iABC platform use
- Usual care (No Intervention): Patients followed in the centers randomized to the control arm will be managed by usual care in accordance with local clinical guidance

INTERVENTIONS:
Other: iABC platform use — The novel platform (iABC) that will be used in AFFIRMO will consist of an educational program, a healthy or functional diet/physical activity, guideline-adherent drug treatments, periodic (re)assessment.
  Arms: Quality-improvement intervention (iABC)

SUMMARY:
The study will verify if a structured multidisciplinary approach (called iABC), aimed to improve the appropriate management of elderly AF patients with multimorbidity (the i-ABC group), would provide a clear evidence of an improvement in clinical conditions and quality of life compared to usual clinical care. The i-ABC group in AFFIRMO will follow the ABC pathway, focused on three domains: avoid stroke with anticoagulation (with optimized VKA or label-adherent DOAC use); better symptom management; and optimized management of associated cardiovascular and non cardiovascular comorbidities.

The study will be conducted in Bulgaria, Denmark, Italy, Romania, Serbia and Spain .

DETAILED DESCRIPTION:
Controlled study, testing a structured implementation of an appropriate management of elderly AF patients with multimorbidity in clinical practice (adapting the ABC pathway and integrating the means of CGA) versus usual care; it is designed to provide reliable evidence of an active holistic integrated management approach to a common, multimorbid and 'high risk' clinical condition.

AFFIRMO use a novel platform (iABC) in a cluster randomized trial design, randomizing centres to iABC versus usual care.

Centres will be selected in each participating country (Bulgaria, Denmark, Italy, Romania, Serbia and Spain) under the responsibility of National Coordinators on the basis of a demonstrated interest in managing patients with AF. The 8-10 participating clusters in each country (see study size below) will be randomized in a 1:1 ratio to receive a quality-improvement intervention (iABC, experimental group) or 'usual care' practice (control group). The randomization will occur in each Country once all clusters selected in the Country have obtained IRB approval. The allocation schedule for random assignment of care models (iABC or usual care) to sites will be computer generated at the Central Coordinating Centre. The clusters in each Country will be stratified in 2 groups: Centres with or without interventional electrophysiology laboratory for AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of both sexes with age ≥65 years;
* First diagnosed, paroxysmal, persistent, long-standing persistent or permanent AF, confirmed as per guideline-recommended diagnostic criteria for AF, e.g. with electrocardiogram (ECG) or Holter monitoring;
* ≥1 additional long-term comorbidity, thus fulfilling the definition of multimorbidity: hypertension (treated with at least 2 antihypertensive drugs), coronary artery disease (CAD), peripheral artery disease, heart failure, stroke/TIA, diabetes mellitus, COPD, CKD.

Exclusion Criteria:

* Mechanical prosthetic heart valve or moderate/severe mitral stenosis;
* Patient unwilling to be enrolled and sign written informed consent;
* Patient unable to understand the study and attend the follow-up;
* Serious diseases with a life expectancy inferior to 12 months;
* Patients included in other interventional studies.

Only for sites randomized to the iABC group:

- Patient without a device suitable for iABC use.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Impact of iABC on all cause unplanned hospitalization | 12 months
  All-cause unplanned hospitalization

SECONDARY OUTCOMES:
Impact of iABC on the composite endpoint of non ischemic stroke, transient ischemic attack and cardiovascular death | 12 months
  A 'composite endpoint' of nonfatal ischemic stroke, transient ischemic attack, and cardiovascular death
Impact of iABC on secondary outcome measures | 12 months
  all-cause mortality
Impact of iABC on secondary outcome measures | 12 months
  all-cause mortality and all-cause (planned and unplanned) hospitalizations
Impact of iABC on secondary outcome measures | 12 months
  new diagnosis of HF or worsening HF requiring hospitalizations
Impact of iABC on secondary outcome measures | 12 months
  quality of life assessed with EQ-5D-5L questionnaire
Impact of iABC on secondary outcome measures | 12 months
  major bleeds defined according to the ISTH definitions
Impact of iABC on secondary outcome measures | 12 months
  intracranial bleeds
Impact of iABC on secondary outcome measures | 12 months
  occurrence of renal dysfunction or worsening renal function
Level of adherence to iABC pathway | 12 months
  Level of adherence to iABC pathway will be evaluated by:
  * the number of accesses to the APP.
  * daily patient's adherence to oral anticoagulant therapy,
  * weekly blood pressure and weight self-measurements input
  * weekly AF symptoms related questionnaires completion
Impact of iABC on self reported physical activity | 12 months
  Impact of iABC on self reported physical activity
Level of empowerment and engagement of patient assessed with PHE-S questionnaire | 12 months
  Level of empowerment and engagement of patient assessed with PHE-S questionnaire
Therapy adherence | 12 months
  Will be evaluated by persistence medical treatment at 12 month follow-up as reported in the e-CRF

CONTACTS AND LOCATIONS:
Locations (50):
- Bulgaria (8):
  - MHAT Haskovo AD-Cardiology, Haskovo
  - SHATS Sveti Georgi - Pernik-Cardiology, Pernik
  - MBAL Sv. Ivan Rilski-Cardiology, Plovdiv
  - UMBAL Sveti Georgi EAD-Clinic of Cardiology, Plovdiv
  - UMHAT Pulmed Plovdiv-Cardiology, Plovdiv
  - Acibadem City Clinic Tokuda Hospital-Dept of Electrophysiology Clinic of Cardiology, Sofia
  - Acibadem City Clinic UMBAL Cardiovascular Center-CARDIOLOGY, Sofia
  - National Heart Hospital-ICCU, Sofia
- Denmark (4):
  - Herlev Hospital-Department of Cardiology, Herlev
  - North Denmark Regional Hospital-Department of Cardiology, Hjørring
  - Horsens Regional Hospital-Department of Medicine, Horsens
  - Silkeborg Regional Hospital-Diagnostic Centre, University Clinic for Development of Innovative Patient Pathways, Silkeborg
- Italy (12):
  - Azienda Ospedaliera S. Anna E S. Sebastiano-Cardiologia Clinica Universitaria, Caserta, CE
  - Ospedale Santa Maria Nuova-Cardiologia - Firenze 1, Florence, FI
  - Als Genovese Palazzo Della Salute-Cardiologia Quarto, Genova, GE
  - Ospedale Della Misericordia-U.O. Di Cardiologia, Grosseto, GR
  - Fondazione Irccs San Gerardo Dei Tintori - Ospedale San Gerardo - U.O.C. Cardiologia, Monza, MB
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Milano-Uo Cure Subacute, Milan, MI
  - Ospedale Civile 'Guglielmo Da Saliceto'-Uoc Cardiologia E Utic, Piacenza, PC
  - Ospedale Gubbio-Gualdo Tadino-U.O. Di Utic E Cardiologia, Gubbio, PG
  - Policlinico Umberto Primo-Medicina Interna E Immunologia Clinica, Roma, RM
  - Azienda Ospedaliera Santa Maria-Medicina Interna, Terni, TR
  - Pou "Santa Maria Della Misericordia"-S.O.C. Cardiologia, Udine, UD
  - Aou Federico Ii-Medicina Metabolico-Riabilitativa, Napoli
- Romania (8):
  - Spitalul Clinic Colentina-Cardiology, Bucharest
  - Spitalul Clinic Colentina-Internal Medicine, Bucharest
  - Spitalul Clinic Coltea-Internal Medicine and Cardiology, Bucharest
  - Spitalul Clinic de Urgenta 'Bagdasar-Arseni'-Cardiology, Bucharest
  - Spitalul Clinic de Urgenta Bucuresti-Cardiology, Bucharest
  - Spitalul Clinic Prof.Dr.Th.Burghele-Internal Medicine and Cardiology, Bucharest
  - Spitalul Universitar de Urgenta Elias-Cardiology, Bucharest
  - Spitalul Universitar de Urgenta Militar Central Dr. Carol Davila-Cardiac Function Laboratory, Bucharest
- Serbia (8):
  - Institute for Cardiovascular Diseases Dedinje-Pacemaker and electrophysiology department, Belgrade
  - KBC Bezanijska Kosa-Cardiology Department, Belgrade
  - KBC Zemun-Cardiology Department, Belgrade
  - University Clinical Centre of Serbia-Department for cardiac arrhythmias, Belgrade
  - University Clinical Centre of Serbia-Department for invasive electrophysiology, Belgrade
  - University Clinical Centre of Serbia-Emergency centre, Belgrade
  - University Clinical Centre of Kragujevac-Cardiology Department, Kragujevac
  - University Clinical Centre of Nis-Cardiology Department, Niš
- Spain (10):
  - Hospital General Universitario de Alicante Doctor Balmis-CARDIOLOGY, Alicante
  - Hospital General Universitario Santa Lucía-CARDIOLOGY, Cartagena
  - Hospital Valle del Guadalhorce-CARDIOLOGY, Cártama
  - Hospital General Universitario de Elche-CARDIOLOGY, Elche
  - Hospital Universitario Virgen de la Victoria-CARDIOLOGY, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca-CARDIOLOGÍA, Murcia
  - Hospital General Universitario Reina Sofía-CARDIOLOGY, Murcia
  - Hospital Universitario San Juan de Alicante-CARDIOLOGY, Sant Joan d'Alacant
  - Hospital Universitario de Tarragona Joan XXIII-Cardiology, Tarragona
  - Pius Hospital de Valls-Cardiology, Valls

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Proietti M, Lip GYH, Ainsworth J, Dan GA, Frost L, Graffigna G, Lucci D, Marin F, Potpara TS, Sanaullah A, Tokmakova M, Johnsen SP, Maggioni AP; AFFIRMO Study Investigators and Consortium. Integrated Care Management for Older Multimorbid Patients with Atrial Fibrillation: Rationale, Design and Baseline Characteristics for the Atrial Fibrillation Integrated Approach in Frail, Multimorbid and Polymedicated Older People (AFFIRMO) trial. Am Heart J. 2026 Jan 22:107356. doi: 10.1016/j.ahj.2026.107356. Online ahead of print. PMID 41580107